CLINICAL TRIAL: NCT03971383
Title: A Multi-Center, Randomized, Double Blind, Placebo-controlled Phase Ⅱc Study of Aolanti Weipang Tablets in Patients With Postprandial Discomfort Syndrome of Functional Dyspepsia to Evaluate the Safety and Validity
Brief Title: Phase Ⅱc Sutdy of Aolanti Weikang Tablets in FD PDS Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QF-WKP-203
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aolanti Weipang Tablets (Experimental): 3 tablets one time, 3 times a day(tid)
  Interventions: Drug: Aolanti Weipang Tablets
- Placebo (Placebo Comparator): 3 tablets one time, 3 times a day(tid)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aolanti Weipang Tablets — 3 tablets one time, 3 times a day(tid)
  Arms: Aolanti Weipang Tablets
Drug: Placebo — 3 tablets one time, 3 times a day(tid)
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and validity of Aolanti Weipang Tablets in Patients with Postprandial Discomfort Syndrome of Functional Dyspepsia

DETAILED DESCRIPTION:
This is a multi-center, randomized, double blind, placebo-controlled phase Ⅱc study to evaluate the safety and validity of Aolanti Weipang Tablets in patients with postprandial discomfort syndrome of Functional Dyspepsia(FD). This study will consecutive about 12 weeks, including 2 weeks of screening, 1 week of blank run-in, 1 week of placebo run-in, 4 weeks of double blind treatment and 4 weeks of observation after treatment. The subjects will be randomly given orally Aolanti Weikang Tablets or placebo tablets at a 1:1 ratio three times a day(tid) with 3 tablets one time for the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with FD according to the ROME Ⅳ criteria，and must with symptom of bothersome postprandial fullness;
* Patients diagnosed with Stagnation of Qi according to traditional Chinese medicine;
* At least the symptom of bothersome postprandial fullness ≥4 on the Visual Analogue Scale(VAS), and the number of recurrence day must ≥3 in one week;
* Provides voluntary informed consent after receiving adequate explanation and demonstrates thorough understanding of the nature of the study.

Exclusion Criteria:

* The patients with high placebo effect, the scores in placebo run-in stage declined much than 30 percent of the mean VAS per week compare to blank run-in stage;
* Unable to take drugs orally;
* Within 7 days of Screening, the average number of stool > 2 times/day;
* Within 7 days of Screening, with the presence of ≥ type 5 stool form per the Bristol Stool Form Scale;
* History of drug or aurantium allergy;
* Patients with positive in fecal occult blood test;
* Abnormal liver and/or kidney function: creatinine >1.5*ULN (upper limits of normal), and/or AST and/or ALT > 2.0*ULN, and/or TBil > 1.5*ULN;
* Patients with family history of prolonged QT syndrome or have history of torsional apical ventricular tachycardia; or QTc > 480 ms;
* Digestive diseases, or other diseases within 6 months before Screening that may affect the swallow, absorption, or metabolism of study drugs, and not yet fully recovered judged by the Investigator;
* Patients who positive in H. Pylori test plan to accept the H. pylori eradication therapy within the trial;
* Serious complications (heart, brain, lung, liver, kidney, or blood disease);
* Neuropsychiatric disorders;
* Use of prohibited medications;
* Pregnant or lactating women or those who are planning to conceive during the study period;
* Drug abuse within 3 months, or alcohol abuse within 6 months;
* Patients participated in other clinical trials within 30 days before taking drugs;
* Other conditions deemed ineligible for enrollment by Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2019-06-10 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-05-03 (Estimated)

PRIMARY OUTCOMES:
The response rate of patient's on the syndrome of postprandial discomfort | 4 weeks
  the response rate of patients on the syndrome of postprandial discomfort, patient's evaluation of symptomatic improvement by overall treatment efficacy is classified by 7 point Likert scale: Significantly improved Improved Slightly improved No change Slightly worse Worse Much worse And only the Improved and Significantly improved classified as responsed.

SECONDARY OUTCOMES:
The response rate of patient's on the syndrome of postprandial discomfort and early satiation | 8 weeks
  the response rate of patient's on the syndrome of postprandial discomfort and early satiation
The response rate of patient's on the syndrome of early satiation | 8 weeks
  the response rate of patient's on the syndrome of early satiation
The safety of Aolanti Weikang Tablets on patients | 8 weeks
  Number and grade of treatment-related adverse events, all of theAE are assessed by NCI-CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Ke, Principal Investigator — The Second People's Hospital of Fujian Province
Locations (1):
- The Second People's Hospital of Fujian Province, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No